CLINICAL TRIAL: NCT04910412
Title: Effects of Transcranial Direct Current Stimulation With Gait Training on Lower Limb Performance in Individual With Incomplete Spinal Cord Injury
Brief Title: Effects of tDCS With Gait Training on Leg Performance in Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 64005
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Incomplete Spinal Cord Injury
Keywords: Transcranial direct current stimulation; Incomplete spinal cord injury; Lower limb performance
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS with gait training (Experimental): Anodal tDCS will be applied over the primary motor cortex (M1) (anodal or active electrode on M1 area, cathodal or reference electrode on supraorbital area) for 20 mins with 2 mA intensity before 50-minute of gait training with external cue and feedback for 5 consecutive sessions
  Interventions: Device: transcranial direct current stimulation
- Sham tDCS with gait training (Active Comparator): Sham tDCS will be applied over the primary motor cortex for 20mins before 50-minute of gait training with external cue and feedback for 5 consecutive sessions
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Transcranial direct current stimulation will be use for the intervention. Anodal and sham tDCS will be applied in 2 mA through a pair of saline-soaked surface sponge electrode 35 cm square for 20 minute over the primary motor area for modulating the cortical excitability before apply the rehabilitation training

SUMMARY:
This study aim to investigate the effects of anodal transcranial direct current stimulation combined with gait training for 5 consecutive session on gait performance, balance, sit to stand performance and quality of life in persons with incomplete SCI at post intervention, 1-month follow-up and 2-month follow up

DETAILED DESCRIPTION:
The result from the previous studies of Water in 1994 regarding the ambulation status of patients with spinal cord injury (SCI) for a period of 1 year after injury. It was found that 76% of incomplete paraplegia and 46 % of incomplete tetraplegia can recovery their walking ability to become community ambulators. However, the recovery rate gradually decreased and started to hit the plateau level around 9 months post injury or in chronic phase. Therefore, it is a challenge in rehabilitation to restore their functions such as walking which is a primary goal of functional independence.

Activity-based rehabilitation therapy (ABRT) (such as locomotion training) is an intensive intervention that has the potential to promote neurological recovery and enhance walking ability in individual with incomplete SCI. Although, ABRT showed positive results in motor function recovery in incomplete SCI survivors, it may not be able to promote full recovery, especially in chronic patients. Recent studies showed that the combination of training with top-down approach may be an option that could promote motor recovery after SCI.

transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that is currently being used as an add-on treatment in neurorehabilitation. tDCS over the primary motor cortex has been shown to modulate neural activity at both cortical and spinal levels. It also produce an after-effect in modulating neuronal synaptic plasticity and increasing the expression of brain-derived neurotrophic factor (BDNF). Early tDCS studies have shown that increasing stimulation intensity or duration within certain limits enhances tDCS efficacy: while anodal stimulation increases cortical excitability, cathodal stimulation decreases it. The application of tDCS is to place the electrode in a specific montage on the decided target brain area and deliver the low-intensity current pass through that brain area for neural modulation during or after providing a rehabilitation program. Previous studies of the application of tDCS showed that applying of tDCS on primary motor cortex with intensity of 2 milliampere (mA) for 10-20 minutes combined with rehabilitation can enhance lower limb performance such as knee strength, ankle movement, and sit to stand performance in people with stroke as well as walking speed in people with Parkinson's disease. According to result from those previous studies can revealed that the combination of rehabilitation with modulation of corticospinal excitability can enhance lower limb performance in individual with neurological condition. In individuals with incomplete SCI, the excitability of the preserved corticospinal pathways is reduced which can affect the control of their motor skills and motor recovery. Several studies reported positive effect of anodal tDCS combined with training in individuals with incomplete SCI, however most of studies focused on upper limb function. Only few studies on the outcome of lower limb function and walking ability, which are required to return to their daily living and thus increase in quality of life (QOL). Moreover, most of studies in the lower limb were conducted in a small sample size and reported inconclusive results.

Therefore, the purpose of this study is to determine whether the effects of combining anodal tDCS with gait training for 5 consecutive session in people with incomplete SCI can improve lower limb performance consist of gait performance(spatiotemporal), dynamic balance(time up and go test), sit to stand performance (5 times of sit to stand test) and QOL after a prolonged period of follow-up at 1-month and 2-month compare to control group of sham tDCS with gait training.

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Injury Association (ASIA) impairment scale C or D
* Age between 18-70 years
* Onset of injury between 1-30 months
* Ability to walk at least 15 meters with or without walking aid

Exclusion Criteria:

* Using other orthoses except the ankle-foot orthosis (AFO)
* Having musculoskeletal pain limiting their walking (pain score > 5/ 10)
* Modified Ashworth Scale (MAS) greater than 2
* Having unstable cardiopulmonary disease
* Having uncontrolled conditions e.g. uncontrolled hypertension, uncontrolled diabetes
* Having a history of other neurological diseases e.g. stroke
* Having contra-indication to use tDCS which are
* The presence of intracranial metal implantation, cochlear implant, or cardiac pacemaker
* Having an open wound or wound infection on the scalp
* Having a history of brain surgery
* Having a history of seizure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in gait efficacy assessed by walking speed(m/s) at 5 days | Baseline and 5 days
  10 meter walk test will be used for measuring walking speed in 2 pace which are 1) comfortable pace 2) fastest safe pace by ask the participants to walk along 14-meter walkway and the assessor will record the time at the middle 10 meters and calculate into speed of walking in m/s. Increasing walking speed indicates better walking performance.
Change from baseline in gait efficacy assessed by walking speed(m/s) at 1 month | Baseline and 1 month
  10 meter walk test will be used for measuring walking speed in 2 pace which are 1) comfortable pace 2) fastest safe pace by ask the participants to walk along 14-meter walkway and the assessor will record the time at the middle 10 meters and calculate into speed of walking in m/s. Increasing walking speed indicates better walking performance.
Change from baseline in gait efficacy assessed by walking speed (m/s) at 2 months | Baseline and 2 months
  10 meter walk test will be used for measuring walking speed in 2 pace which are 1) comfortable pace 2) fastest safe pace by ask the participants to walk along 14-meter walkway and the assessor will record the time at the middle 10 meters and calculate into speed of walking in m/s. Increasing walking speed indicates better walking performance.

SECONDARY OUTCOMES:
Change from baseline in gait efficacy assessed by stride parameter (m) at 5 days | Baseline and 5 days
  G walk accelerometer will be use for measuring stride component of walking with comfortable pace. The assessor will attach the device with belt at L5 spinous process and ask the participants to walk with their comfortable pace and record the parameter then transfer to computer. The increasing of stride length indicates good walking performance. The reducing of stride duration indicates good walking performance.
Change from baseline in gait efficacy assessed by stride parameter (m) at 1 month | Baseline and 1 month
  G walk accelerometer will be use for measuring stride component of walking with comfortable pace. The assessor will attach the device with belt at L5 spinous process and ask the participants to walk with their comfortable pace and record the parameter then transfer to computer. The increasing of stride length indicates good walking performance. The reducing of stride duration indicates good walking performance.
Change from baseline in gait efficacy assessed by stride parameter (m) at 2 months | Baseline and 2 months
  G walk accelerometer will be use for measuring stride component of walking with comfortable pace. The assessor will attach the device with belt at L5 spinous process and ask the participants to walk with their comfortable pace and record the parameter then transfer to computer. The increasing of stride length indicates walking performance. The reducing of stride duration indicates walking performance.
Change from baseline in gait efficacy assessed by cadence (step/min) at 5 days | Baseline and 5 days
  G walk accelerometer will be use for measuring cadence of walking with comfortable pace. The assessor will attach the device with belt at L5 spinous process and ask the participants to walk with their comfortable pace and record the parameter then transfer to computer. The increasing of cadence indicates good walking performance.
Change from baseline in gait efficacy assessed by cadence (step/min) at 1 month | Baseline and 1 month
  G walk accelerometer will be use for measuring cadence of walking with comfortable pace. The assessor will attach the device with belt at L5 spinous process and ask the participants to walk with their comfortable pace and record the parameter then transfer to computer. The increasing of cadence indicates good walking performance.
Change from baseline in gait efficacy assessed by cadence (step/min) at 2 months | Baseline and 2 months
  G walk accelerometer will be use for measuring cadence of walking with comfortable pace. The assessor will attach the device with belt at L5 spinous process and ask the participants to walk with their comfortable pace and record the parameter then transfer to computer. The increasing of cadence indicates good walking performance.
Change from baseline in balance efficacy assessed by duration of timed up and go test at 5 days | Baseline and 5 days
  The timed up and go test will used for assessing dynamic balance of participants by asking the participant to stand up from standard chair with back rest and walk forward for 3 meters and return to sit down at the chair again. The assessor will record the time spending when instructing the participants to start and stop record time when the participants sit down and back against the back rest again. The shorter time indicates good dynamic balance.
Change from baseline in balance efficacy assessed by duration of timed up and go test (s) at 1 month | Baseline and 1 month
  The timed up and go test will used for assessing dynamic balance of participants by asking the participant to stand up from standard chair with back rest and walk forward for 3 meters and return to sit down at the chair again. The assessor will record the time spending when instructing the participants to start and stop record time when the participants sit down and back against the back rest again. The shorter time indicates good dynamic balance.
Change from baseline in balance efficacy assessed by duration of timed up and go test (s) at 2 months | Baseline and 2 months
  The timed up and go test will used for assessing dynamic balance of participants by asking the participant to stand up from standard chair with back rest and walk forward for 3 meters and return to sit down at the chair again. The assessor will record the time spending when instructing the participants to start and stop record time when the participants sit down and back against the back rest again. The shorter time indicates good dynamic balance.
Change from baseline in balance efficacy assessed by duration of five time sit to stand test (s) at 5 days | Baseline and 5 days
  Five time sit to stand test will be used for measuring leg strength and dynamic balance. The assessor will ask the participants to standing up from armless chair with back rest for 5 times in a raw as fast as possible. the assessor will record the time spending of complete 5 time of sit to stand that start from giving instruction and stop when the participant completely sit on chair at 5th repetition. The shorter time indicates good performance
Change from baseline in balance efficacy assessed by duration of five time sit to stand test(s) at 1 month | Baseline and 1 month
  Five time sit to stand test will be used for measuring leg strength and dynamic balance. The assessor will ask the participants to standing up from armless chair with back rest for 5 times in a raw as fast as possible. the assessor will record the time spending of complete 5 time of sit to stand that start from giving instruction and stop when the participant completely sit on chair at 5th repetition. The shorter time indicates good performance
Change from baseline in balance efficacy assessed by duration of five time sit to stand test (s) at 2 months | Baseline and 2 months
  Five time sit to stand test will be used for measuring leg strength and dynamic balance. The assessor will ask the participants to standing up from armless chair with back rest for 5 times in a raw as fast as possible. the assessor will record the time spending of complete 5 time of sit to stand that start from giving instruction and stop when the participant completely sit on chair at 5th repetition. The shorter time indicates good performance
Change from baseline in quality of life assessed by WHOQOL-Bref Thai version (score 26-130) at 1 month | Baseline and 1 month
  World Health Organization (WHO) quality of life (QOL)- bref Thai version will be use for assessing in quality of life. there are two types of questions which are the perceived objective and the self-report subjective and consist of four components of well-being which are physical, psychological, social, and environmental. Each item will be scored from 1-5. (Total score 26-130). The higher score indicates better QOL.
Change from baseline in quality of life assessed by WHOQOL-Bref Thai version (score 26-130) at 2 months | Baseline and 2 month
  WHO quality of life (QOL)- bref Thai version will be use for assessing in quality of life. there are two types of questions which are the perceived objective and the self-report subjective and consist of four components of well-being which are physical, psychological, social, and environmental. Each item will be scored from 1-5 (Total score 26-130). The higher score indicates better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Study Director — Mahidol University
Locations (1):
- Sirindhorn National Medical Rehabilitation Institute, Nonthaburi, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klamruen P, Suttiwong J, Aneksan B, Muangngoen M, Denduang C, Klomjai W. Effects of Anodal Transcranial Direct Current Stimulation With Overground Gait Training on Lower Limb Performance in Individuals With Incomplete Spinal Cord Injury. Arch Phys Med Rehabil. 2024 May;105(5):857-867. doi: 10.1016/j.apmr.2023.09.025. Epub 2023 Nov 4. PMID 37926224